CLINICAL TRIAL: NCT00930098
Title: A Phase II, Open-Label Study of Clofarabine in Paediatric Patients With Refractory/Relapsed Acute Lymphoblastic Leukaemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Bioenvision (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOV-111; UKCCSG: NAG 2003 06
Record Dates: First submitted 2009-06-17; First posted 2009-06-30 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; clolar; evoltra; clofarabine; refractory/relapsed acute leukemia; pediatric acute leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: clofarabine
  Other Names: US Tradename = Clolar; EU Tradename = Evoltra

SUMMARY:
This study is for a population of patients with few or no alternative options that was conducted to determine the response rate to clofarabine. Additionally the study will provide information on the safety profile, impact of overall survival, and impact on remission duration with clofarabine. It is a single arm study and has no comparator.

DETAILED DESCRIPTION:
Note: This clinical trial was conducted by Bioenvision Ltd. Bioenvision Ltd. was acquired by Genzyme Corporation Oct 2007.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of ALL and confirmed by pathologic assessment.
* Be ≤ 21 years old at time of initial diagnosis.
* Eligible patients must have: Primary refractory disease; OR relapsed or refractory disease after a minimum of 2 prior blocks of treatment.
* Must not be eligible for therapy of higher curative potential.
* Have a Karnofsky Performance Status of ≥ 50 or Lansky Performance Scale of ≥ 30.
* Provide a signed, written informed consent from parent or guardian or young adult patients.
* Be able to comply with study procedures and follow-up examinations.
* Have adequate cardiac function without treatment.
* Have adequate organ function as indicated by the laboratory values for serum creatinine, serum bilirubin, AST and ALT, obtained within 7 days prior to registration.

Exclusion Criteria:

* Received previous treatment with clofarabine.
* Patients with isolated extramedullary disease.
* Have received prior BMT or PBSCT within the last 6 months.
* Have received prior BMT or PBSCT more than 6 months ago, but now has compromised organ function.
* Have an active, uncontrolled systemic infection.
* Are pregnant or lactating. Male and female patients who are fertile must agree to use an effective means of birth control to avoid pregnancy.
* Have a psychiatric disorder that would interfere with consent, study participation, or follow-up.
* Have received any other chemotherapy within the previous 2 weeks and must have recovered from acute toxicity oa all previous therapy prior to enrollment.
* Have any other severe concurrent disease.
* Have recent history of significant renal, hepatic or pulmonary dysfunction, or cardiac dysfunction or on treatment to support cardiac function.
* Have CNS disease.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2003-12; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate after 1 course or more | minimum of 1 course and maximum of 12 courses

SECONDARY OUTCOMES:
Overall response rate after 2 courses or more | minimum of 2 courses and maximum of 12 courses
Rate of response (complete, complete with incomplete blood count recovery, partial) after 1 course or more | minimum of 1 course and maximum of 12 courses
Time-to-event parameters including duration of remission and overall survival | Until death of patient or until end of study treatment for last enrolled patient
Safety and tolerability | Until death of patient or until end of study treatment for last enrolled patient
Number of patients received bone marrow or peripheral blood stem cell transplantation and the time to transplant following commencement of Clofarabine | Until death of patient or until end of study treatment for last enrolled patient
Determine pharmacokinetic profile and intracellular triphosphate and levels of clofarabine | every day during the first course of treatment
Document the metabolic pathways that may predict Clofarabine sensitivity or resistance | day 1, day 5, day 6 and day 7 of the first course

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (36):
- Vienna, Austria
- France (9):
  - Besançon
  - Bordeaux
  - Lille
  - Lyon
  - Marseille
  - Nantes
  - Paris
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (9):
  - Berlin
  - Düsseldorf
  - Frankfurt
  - Hamburg
  - Hanover
  - Kiel
  - Munich
  - Münster
  - Stuttgart
- Italy (2):
  - Monza
  - Pavia
- Netherlands (5):
  - Amsterdam
  - Groningen
  - Leiden
  - Rotterdam
  - Utrecht
- United Kingdom (10):
  - Birmingham
  - Bristol
  - Glasgow
  - Leeds
  - Liverpool
  - London
  - Manchester
  - Newcastle upon Tyne
  - Sheffield
  - Sutton